CLINICAL TRIAL: NCT00637000
Title: Induction of Opioid-Dependent Individuals Onto Buprenorphine and Buprenorphine/Naloxone
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Indivior Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RB-US-07-0002
Record Dates: First submitted 2008-03-10; First posted 2008-03-17 (Estimated); Results first posted 2014-05-09 (Estimated); Last update posted 2017-06-05 (Actual); Status verified 2017-04

CONDITIONS: Opioid-related Disorders
Keywords: Opioid dependence; Opioid withdrawal symptoms
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Buprenorphine; Buprenorphine, Naloxone Drug Combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Buprenorphine soluble film (Experimental): Day 1: Buprenorphine soluble film administered at a dose of 4 mg 3 times per day, plus placebo. Dosing occurred at 0900, 1100, and 2000 hours.
  Days 2-5: Buprenorphine soluble film administered at a dose of 16 mg to 24 mg once per day, plus placebo. Dosing occurred at 0900 hours.
  Interventions: Drug: Buprenorphine soluble film; Drug: Placebo
- Buprenorphine/naloxone soluble film (Experimental): Day 1: Buprenorphine/naloxone soluble film administered at a dose of 4mg/1mg 3 times per day, plus placebo. Dosing occurred at 0900, 1100, and 2000 hours.
  Days 2 to 5: Buprenorphine/naloxone soluble film administered at a dose of 16mg/4 mg to 24 mg/6 mg once per day, plus placebo. Dosing occurred at 0900 hours.
  Interventions: Drug: Buprenorphine/naloxone film strip; Drug: Placebo

INTERVENTIONS:
Drug: Buprenorphine soluble film — Buprenorphine soluble film strips administered sublingually with doses escalated from 12 mg per day up to 24 mg daily for 5 days of total treatment.
  Other Names: Subutex
  Arms: Buprenorphine soluble film
Drug: Buprenorphine/naloxone film strip — Buprenorphine/naloxone soluble film strips administered sublingually with doses escalated from 12 mg buprenorphine/3 mg naloxone to 24 mg buprenorphine /6 mg naloxone daily for 5 days of total treatment.
  Other Names: Suboxone
  Arms: Buprenorphine/naloxone soluble film
Drug: Placebo — Placebo soluble film administered on the same schedule as active treatment to maintain the study blind.

SUMMARY:
The purpose of this study is to compare the presence, degree, time course and profile of opioid withdrawal symptoms associated with induction onto new formulations of buprenorphine or buprenorphine/naloxone in persons with active opioid dependence. The primary outcome measure is the severity of withdrawal symptoms measured using the Clinical Opiate Withdrawal Scale (COWS). The primary study hypothesis is that neither drug formulation will precipitate an opioid withdrawal syndrome.

DETAILED DESCRIPTION:
Buprenorphine sublingual and buccal soluble films are being developed to be used for the same indication and over the same buprenorphine dose range as Subutex and Suboxone sublingual tablets in the treatment of opioid dependence. However, only films administered by the sublingual route were evaluated in this study.

The soluble film dosage is expected to provide the following enhancements and potential advantages over the current Subutex and Suboxone product:

* Mitigation against unintentional pediatric exposure by providing child-resistant packaging in unit dose format.
* Improvement in subject convenience and compliance by ensuring rapid disintegration.
* Protection against diversion by providing a dosage form that is very difficult for the subject to remove from the sublingual or buccal mucosa after administration. This provides assurance to the caregiver that the dose has actually been taken appropriately in a supervised setting.
* Provision of a unit dose product format for hospital and institutional use.
* Decreased product damage during shipping as compared to Subutex and Suboxone tablets.

ELIGIBILITY:
Inclusion Criteria:

Subject must:

* Provide written informed consent.
* Have a Diagnostic and Statistical Manual of Mental Disorders-IV (DSM-IV) diagnosis of opioid dependence.
* Be male or female, 18 to 65 years of age, inclusive.
* If female, have a negative pregnancy test during screening and agree to use an acceptable method of birth control.

Exclusion Criteria:

Subjects must not:

* Have participated in an experimental drug or device study within the last 30 days.
* Be currently (past 30 days from start of screening) engaged in opioid agonist, opioid partial agonist, or opioid antagonist treatment.
* If female, be breast feeding or lactating.
* Have any medical condition that in the opinion of the physician investigator would preclude the subject from completing the study.
* Have any clinically significant non-substance use psychiatric disorder (e.g., schizophrenia).
* Have current suicidal ideation.
* Have a Mini Mental Status Exam score less than 24.
* Have physical dependence on alcohol.
* Have physical dependence on sedative-hypnotics.
* Have active aphthous stomatitis.
* Have active oral herpes.
* Need on-going prescription medications that interact with the P450 3A4 (a member of the cytochrome P450 superfamily of enzymes) system.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2008-03; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric C. Strain, M.D., Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University School of Medicine, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patient enrollment commenced 03/19/08 and was completed 09/19/08. The study site was an in-patient research-based clinic affiliated with Johns Hopkins University School of Medicine.
Pre-assignment Details: During screening run-in, subjects received 30 mg morphine subcutaneously up to 4 times/day for up to 13 days. Subjects underwent two test sessions, consisting of a challenge of naloxone (0.4 mg) or placebo intramuscularly and evaluation for the severity of withdrawal. Subjects able to detect withdrawal were randomized to treatment.
Groups:
- Sublingual Buprenorphine Soluble Film: Day 1: Buprenorphine soluble film administered at a dose of 4 mg 3 times per day, plus placebo. Dosing occurred at 0900, 1100, and 2000 hours.
  Days 2-5: Buprenorphine soluble film administered at a dose of 16 mg to 24 mg once per day, plus placebo. Dosing occurred at 0900 hours.
- Sublingual Buprenorphine/Naloxone Soluble Film: Day 1: Buprenorphine/naloxone soluble film administered at a dose of 4mg/1mg 3 times per day, plus placebo. Dosing occurred at 0900, 1100, and 2000 hours.
  Days 2 to 5: Buprenorphine/naloxone soluble film administered at a dose of 16mg/4 mg to 24 mg/6 mg once per day, plus placebo. Dosing occurred at 0900 hours.
Period: Overall Study
Arm/Group | Sublingual Buprenorphine Soluble Film | Sublingual Buprenorphine/Naloxone Soluble Film
Started | 20 (Randomized and treated) | 18 (Randomized and treated)
Evaluable | 18 | 16
Completed | 16 | 15
Not Completed | 4 | 3
Not completed — Withdrawal by Subject | 4 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sublingual Buprenorphine Soluble Film | Sublingual Buprenorphine/Naloxone Soluble Film | Total
Number analyzed (Participants) | 20 | 18 | 38
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 18 | 38
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.2 (10) | 40.2 (7.9) | 40.2 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 7 | 12
  Male | 15 | 11 | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 20 | 18 | 38
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 8 | 4 | 12
  White | 12 | 13 | 25
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 20 | 18 | 38

OUTCOME MEASURES:

1. Primary Outcome: Severity of Withdrawal Symptoms Measured Using the Clinical Opiate Withdrawal Scale (COWS) at Baseline and the Peak COWS up to 23.5 Hours After the First Administration
Description: The COWS is an 11-item instrument used to assess symptoms of opioid withdrawal (Wesson et al., 1999). The score is the sum of the response to each of the 11 items and cover a range of 0-48. The COWS is commonly used by clinicians treating patients with buprenorphine to monitor the severity of withdrawal. COWS scores below 5 are considered not indicative of withdrawal. Scores from 5 to 12 are considered mild withdrawal; from 13 to 24 moderate withdrawal; 25 to 36 moderate/severe withdrawal, and 37-48 severe withdrawal.
  The baseline COWS was the score obtained 30 minutes prior to administration of soluble films on Day 1. Peak COWS was the highest COWS score obtained between 1-23.5 hours post administration on Day 1.
Time Frame: Baseline: 30 minutes prior to first administration on Day 1. Peak: up to 23.5 hours post administration on Day 1
Population: Per protocol, the evaluable population includes all subjects randomized to the study who completed the study through the first two days of soluble films administration and assessments for 23.5 hours after the first day of soluble films administration.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sublingual Buprenorphine Soluble Film | Sublingual Buprenorphine/Naloxone Soluble Film
Number analyzed (Participants) | 18 | 16
units on a scale
  Baseline | 9.1 (5.5) | 10.1 (6.4)
  Peak | 4.2 (2.4) | 5.7 (3.2)
Statistical Analysis 1: Comparison: Sublingual Buprenorphine Soluble Film vs Sublingual Buprenorphine/Naloxone Soluble Film; To test the primary study hypothesis that neither soluble film formulation would precipitate an opioid withdrawal syndrome, peak COWS score in the 23.5 hour period after the initial soluble film administration were compared to pre-administration baseline COWS scores (30 minutes prior to soluble film administration) using a group by time repeated measures model with a first-order autoregressive covariance structure; Test type: Superiority or Other; p < 0.0001, Repeated measures model — The p-value was not adjusted for multiple comparisons; The statistical method used was a group by time repeated measures model with a first-order autoregressive covariance structure

2. Secondary Outcome: Severity of Withdrawal Symptoms Measured Using the Clinical Opiate Withdrawal Scale (COWS) at the End of Induction and the Peak COWS Post Induction
Description: The COWS is an 11-item instrument used to assess symptoms of opioid withdrawal (Wesson et al., 1999). The score is the sum of the response to each of the 11 items and cover a range of 0-48. The COWS is commonly used by clinicians treating patients with buprenorphine to monitor the severity of withdrawal. COWS scores below 5 are considered not indicative of withdrawal. Scores from 5 to 12 are considered mild withdrawal; from 13 to 24 moderate withdrawal; 25 to 36 moderate/severe withdrawal, and 37-48 severe withdrawal.
  The end of induction COWS was the score obtained 47.5 hours after first administration of soluble films on Day 1. Peak post induction COWS was the highest COWS score obtained on Days 2-5.
Time Frame: End of Induction: 47.5 hours after first administration Peak Post Induction: Days 3-5
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sublingual Buprenorphine Soluble Film | Sublingual Buprenorphine/Naloxone Soluble Film
Number analyzed (Participants) | 18 | 16
units on a scale
  End of Induction | 0.6 (0.5) | 1.0 (1.0)
  Peak Post Induction | 1.0 (1.0) | 2.6 (2.4)
Statistical Analysis 1: Comparison: Sublingual Buprenorphine Soluble Film vs Sublingual Buprenorphine/Naloxone Soluble Film; Test type: Superiority or Other; p = 0.000, Repeated measures model; Group by time repeated measures model with a first-order autoregressive covariance structure

3. Secondary Outcome: Pupil Diameter Measurements at Baseline and the Maximum Pupil Diameter up to 23.5 Hours After the First Administration
Description: Pupil diameter was measured at baseline and at intervals post drug administration on Day 1. Peak measurement is the maximum pupil diameter recorded from 15 minutes to 23.5 hours post administration of study intervention.
Time Frame: Baseline: 15 minutes prior to first administration on Day 1. Peak: 15 minutes - 23.5 hours post administration on Day 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Sublingual Buprenorphine Soluble Film | Sublingual Buprenorphine/Naloxone Soluble Film
Number analyzed (Participants) | 18 | 16
mm
  Baseline | 6.24 (0.97) | 6.11 (0.88)
  Peak | 4.39 (6.27) | 5.99 (0.98)
Statistical Analysis 1: Comparison: Sublingual Buprenorphine Soluble Film vs Sublingual Buprenorphine/Naloxone Soluble Film; Test type: Superiority or Other; p = 0.035, Repeated measures model — The p-value was not adjusted for multiple comparisons; Group by time repeated measures model with a first-order autoregressive covariance structure

4. Secondary Outcome: Pupil Diameter Measurements at Baseline and the Minimum Pupil Diameter up to 23.5 Hours After the First Administration
Description: Pupil diameter was measured at baseline and at intervals post drug administration on Day 1. Peak measurement is the minimum pupil diameter recorded from 15 minutes to 23.5 hours post administration of study intervention.
Time Frame: Baseline: 15 minutes prior to first administration on Day 1. Peak: 15 minutes - 23.5 hours post administration on Day 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Sublingual Buprenorphine Soluble Film | Sublingual Buprenorphine/Naloxone Soluble Film
Number analyzed (Participants) | 18 | 16
mm
  Baseline | 6.24 (0.97) | 6.11 (0.88)
  Peak | 4.39 (1.27) | 4.32 (1.08)
Statistical Analysis 1: Comparison: Sublingual Buprenorphine Soluble Film vs Sublingual Buprenorphine/Naloxone Soluble Film; Test type: Superiority or Other; p < 0.0001, Repeated measures model; Group by time repeated measures model with a first-order autoregressive covariance structure

5. Secondary Outcome: Pupil Diameter Measurements At End of Induction (End of Day 2) and the Minimum Pupil Diameter During the Post Induction Period (Days 3-5)
Description: Pupil diameter was measured at the end of induction (47.5 hours after the first administration of study intervention) and at intervals during the post-induction period (Days 3-5). Peak post induction measurement is the minimum pupil diameter recorded during days 3-5.
Time Frame: End of Induction: 47.5 hours after first administration Peak Post Induction: Days 3-5
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Sublingual Buprenorphine Soluble Film | Sublingual Buprenorphine/Naloxone Soluble Film
Number analyzed (Participants) | 18 | 16
mm
  End of Induction | 5.3 (1.2) | 5.1 (1.2)
  Peak Post Induction | 4.1 (1.1) | 3.6 (0.9)
Statistical Analysis 1: Comparison: Sublingual Buprenorphine Soluble Film vs Sublingual Buprenorphine/Naloxone Soluble Film; Test type: Superiority or Other; p < 0.0001, Repeated measures model; Group by time repeated measures model with a first-order autoregressive covariance structure

6. Secondary Outcome: Visual Analog Scale (VAS) Score at Baseline and the Peak (Maximum Increase) VAS up to 23.5 Hours After First Administration for the Question: "How High Are You?"
Description: A visual analog scale (VAS) was used by participants to answer the subjective question, "How high are you?". The question was one of six used to measure the extent of opioid blockade following study intervention. VAS questions were selected based on previous demonstration of their sensitivity to opioid agonist and antagonist effects (Preston et al., 1988). Participants indicated how high they feel by marking a score on a horizontal line with 0=not high and 100=extremely high.
  The baseline VAS was the score obtained 30 minutes prior to administration of soluble films on Day 1. Peak VAS was the highest VAS score obtained between 1-23.5 hours post administration on Day 1.
Time Frame: Baseline: 30 minutes prior to first administration on Day 1. Peak: up to 23.5 hours post administration on Day 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sublingual Buprenorphine Soluble Film | Sublingual Buprenorphine/Naloxone Soluble Film
Number analyzed (Participants) | 18 | 16
units on a scale
  Baseline | 0.0 (0.0) | 0.0 (0.3)
  Peak | 5.8 (12.9) | 13.7 (24.0)
Statistical Analysis 1: Comparison: Sublingual Buprenorphine Soluble Film vs Sublingual Buprenorphine/Naloxone Soluble Film; Test type: Superiority or Other; p = 0.006, Repeated measures model — The p-value was not adjusted for multiple comparisons; Group by time repeated measures model with a first-order autoregressive covariance structure

7. Secondary Outcome: Visual Analog Scale (VAS) Score at Baseline and the Peak (Maximum Increase) VAS up to 23.5 Hours After First Administration for the Question: "Do You Feel Any Drug Effect?"
Description: A visual analog scale (VAS) was used by participants to answer the subjective question, "Do you feel any drug effect?". The question was one of six used to measure the extent of opioid blockade following study intervention. VAS questions were selected based on previous demonstration of their sensitivity to opioid agonist and antagonist effects (Preston et al., 1988). Participants indicated how high they feel by marking a score on a horizontal line with 0=no effect and 100=maximum effect.
Time Frame: Baseline: 30 minutes prior to first administration on Day 1. Peak: up to 23.5 hours post administration on Day 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sublingual Buprenorphine Soluble Film | Sublingual Buprenorphine/Naloxone Soluble Film
Number analyzed (Participants) | 18 | 16
units on a scale
  Baseline | 0.0 (0.0) | 0.0 (0.0)
  Peak | 44.3 (31.5) | 50.4 (26.0)
Statistical Analysis 1: Comparison: Sublingual Buprenorphine Soluble Film vs Sublingual Buprenorphine/Naloxone Soluble Film; Test type: Superiority or Other; p < 0.0001, Repeated measures model — The p-value was not adjusted for multiple comparisons; Group by time repeated measures model with a first-order autoregressive covariance structure

8. Secondary Outcome: Visual Analog Scale (VAS) Score at Baseline and the Peak (Maximum Increase) VAS up to 23.5 Hours After First Administration for the Question: "Does the Drug Have Any Good Effects?"
Description: A visual analog scale (VAS) was used by participants to answer the subjective question, "Do you feel any good effects?". The question was one of six used to measure the extent of opioid blockade following study intervention. VAS questions were selected based on previous demonstration of their sensitivity to opioid agonist and antagonist effects (Preston et al., 1988). Participants indicated how high they feel by marking a score on a horizontal line with 0=no good effects and 100=maximum good effects.
Time Frame: Baseline: 30 minutes prior to first administration on Day 1. Peak: up to 23.5 hours post administration on Day 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sublingual Buprenorphine Soluble Film | Sublingual Buprenorphine/Naloxone Soluble Film
Number analyzed (Participants) | 18 | 16
units on a scale
  Baseline | 0.0 (0.0) | 0.0 (0.0)
  Peak | 62.3 (35.1) | 57.6 (31.4)
Statistical Analysis 1: Comparison: Sublingual Buprenorphine Soluble Film vs Sublingual Buprenorphine/Naloxone Soluble Film; Test type: Superiority or Other; p < 0.0001, Repeated measures model — The p-value was not adjusted for multiple comparisons; Group by time repeated measures model with a first-order autoregressive covariance structure

9. Secondary Outcome: Visual Analog Scale (VAS) Score at Baseline and the Peak (Maximum Increase) VAS up to 23.5 Hours After First Administration for the Question: "Does the Drug Have Any Bad Effects?"
Description: A visual analog scale (VAS) was used by participants to answer the subjective question, "Does the drug have any bad effects?". The question was one of six used to measure the extent of opioid blockade following study intervention. VAS questions were selected based on previous demonstration of their sensitivity to opioid agonist and antagonist effects (Preston et al., 1988). Participants indicated how high they feel by marking a score on a horizontal line with 0=no bad effects and 100=maximum bad effects.
Time Frame: Baseline: 30 minutes prior to first administration on Day 1. Peak: up to 23.5 hours post administration on Day 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sublingual Buprenorphine Soluble Film | Sublingual Buprenorphine/Naloxone Soluble Film
Number analyzed (Participants) | 18 | 16
units on a scale
  Baseline | 0.0 (0.0) | 12.5 (34.2)
  Peak | 4.4 (11.8) | 6.1 (12.5)
Statistical Analysis 1: Comparison: Sublingual Buprenorphine Soluble Film vs Sublingual Buprenorphine/Naloxone Soluble Film; Test type: Superiority or Other; p = 0.762, Repeated measures model — The p-value was not adjusted for multiple comparisons; Group by time repeated measures model with a first-order autoregressive covariance structure

10. Secondary Outcome: CVisual Analog Scale (VAS) Score at Baseline and the Peak (Maximum Increase) VAS up to 23.5 Hours After First Administration for the Question: "Do You Like the Drug?"
Description: A visual analog scale (VAS) was used by participants to answer the subjective question, "Do you like the drug?". The question was one of six used to measure the extent of opioid blockade following study intervention. VAS questions were selected based on previous demonstration of their sensitivity to opioid agonist and antagonist effects (Preston et al., 1988). Participants indicated how high they feel by marking a score on a horizontal line with 0=no liking and 100=maximum liking.
Time Frame: Baseline: 30 minutes prior to first administration on Day 1. Peak: up to 23.5 hours post administration on Day 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sublingual Buprenorphine Soluble Film | Sublingual Buprenorphine/Naloxone Soluble Film
Number analyzed (Participants) | 18 | 16
units on a scale
  Baseline | 0.0 (0.0) | 0.0 (0.0)
  Peak | 61.2 (40.0) | 59.4 (34.1)
Statistical Analysis 1: Comparison: Sublingual Buprenorphine Soluble Film vs Sublingual Buprenorphine/Naloxone Soluble Film; Test type: Superiority or Other; p < 0.0001, Repeated measures model — The p-value was not adjusted for multiple comparisons; Group by time repeated measures model with a first-order autoregressive covariance structure

11. Secondary Outcome: Visual Analog Scale (VAS) Score at Baseline and the Peak (Maximum Increase) VAS up to 23.5 Hours After First Administration for the Question: "Does the Drug Make You Sick?"
Description: A visual analog scale (VAS) was used by participants to answer the subjective question, "Does the drug make you sick?". The question was one of six used to measure the extent of opioid blockade following study intervention. VAS questions were selected based on previous demonstration of their sensitivity to opioid agonist and antagonist effects (Preston et al., 1988). Participants indicated how high they feel by marking a score on a horizontal line with 0=no effect and 100=maximum effect.
Time Frame: Baseline: 30 minutes prior to first administration on Day 1. Peak: up to 23.5 hours post administration on Day 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sublingual Buprenorphine Soluble Film | Sublingual Buprenorphine/Naloxone Soluble Film
Number analyzed (Participants) | 18 | 16
units on a scale
  Baseline | 0.0 (0.0) | 12.5 (34.2)
  Peak | 2.1 (6.1) | 4.5 (12.3)
Statistical Analysis 1: Comparison: Sublingual Buprenorphine Soluble Film vs Sublingual Buprenorphine/Naloxone Soluble Film; Test type: Superiority or Other; p = 0.349, Repeated measures model — The p-value is not adjusted for multiple comparisons; Group by time repeated measures model with a first-order autoregressive covariance structure

12. Secondary Outcome: Visual Analog Scale (VAS) Scores at End of Induction Period and the Post-induction Period (Maximum Increase) for the Question: "How High Are You?"
Description: A visual analog scale (VAS) was used by participants to answer the subjective question, "How high are you?". The question was one of six used to measure the extent of opioid blockade following study intervention. VAS questions were selected based on previous demonstration of their sensitivity to opioid agonist and antagonist effects (Preston et al., 1988). Participants indicated how high they feel by marking a score on a horizontal line with 0=not high and 100=extremely high.
Time Frame: End of Induction: 47.5 hours after first administration Peak Post Induction: Days 3-5
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sublingual Buprenorphine Soluble Film | Sublingual Buprenorphine/Naloxone Soluble Film
Number analyzed (Participants) | 18 | 16
units on a scale
  End of Induction | 0.0 (0.0) | 6.3 (25.0)
  Peak Post Induction | 8.2 (18.2) | 12.9 (30.1)
Statistical Analysis 1: Comparison: Sublingual Buprenorphine Soluble Film vs Sublingual Buprenorphine/Naloxone Soluble Film; Test type: Superiority or Other; p = 0.028, Repeated measures model — The p-value was not adjusted for multiple comparisons; Group by time repeated measures model with a first-order autoregressive covariance structure

13. Secondary Outcome: Visual Analog Scale (VAS) Scores at End of Induction Period and the Post-induction Period (Maximum Increase) for the Question: "Do You Feel Any Drug Effect?"
Description: as for outcome 7
Time Frame: End of Induction: 47.5 hours after first administration Peak Post Induction: Days 3-5
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sublingual Buprenorphine Soluble Film | Sublingual Buprenorphine/Naloxone Soluble Film
Number analyzed (Participants) | 18 | 16
units on a scale
  End of Induction | 7.9 (16.8) | 15.9 (28.6)
  Peak Post Induction | 53.2 (41.0) | 47.4 (27.8)
Statistical Analysis 1: Comparison: Sublingual Buprenorphine Soluble Film vs Sublingual Buprenorphine/Naloxone Soluble Film; Test type: Superiority or Other; p < 0.0001, Repeated measures model — The p-value was not adjusted for multiple comparisons; Group by time repeated measures model with a first-order autoregressive covariance structure

14. Secondary Outcome: Visual Analog Scale (VAS) Scores at End of Induction Period and the Post-induction Period (Maximum Increase) for the Question: "Do You Feel Any Good Effects?"
Description: as for outcome 8
Time Frame: End of Induction: 47.5 hours after first administration Peak Post Induction: Days 3-5
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sublingual Buprenorphine Soluble Film | Sublingual Buprenorphine/Naloxone Soluble Film
Number analyzed (Participants) | 18 | 16
units on a scale
  End of Induction | 11.0 (26.0) | 20.2 (30.0)
  Peak Post Induction | 61.7 (39.8) | 52.9 (33.1)
Statistical Analysis 1: Comparison: Sublingual Buprenorphine Soluble Film vs Sublingual Buprenorphine/Naloxone Soluble Film; Test type: Superiority or Other; p < 0.0001, Repeated measures model — The p-value was not adjusted for multiple comparisons; Group by time repeated measures model with a first-order autoregressive covariance structure

15. Secondary Outcome: Visual Analog Scale (VAS) Scores at End of Induction Period and the Post-induction Period (Maximum Increase) for the Question: "Does the Drug Have Any Bad Effects?"
Description: as for outcome 9
Time Frame: End of Induction: 47.5 hours after first administration Peak Post Induction: Days 3-5
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sublingual Buprenorphine Soluble Film | Sublingual Buprenorphine/Naloxone Soluble Film
Number analyzed (Participants) | 18 | 16
units on a scale
  End of Induction | 0.0 (0.0) | 0.3 (0.8)
  Peak Post Induction | 0.4 (1.2) | 0.4 (1.2)
Statistical Analysis 1: Comparison: Sublingual Buprenorphine Soluble Film vs Sublingual Buprenorphine/Naloxone Soluble Film; Test type: Superiority or Other; p = 0.117, Repeated measures model — The p-value was not adjusted for multiple comparisons; Group by time repeated measures model with a first-order autoregressive covariance structure

16. Secondary Outcome: Visual Analog Scale (VAS) Scores at End of Induction Period and the Post-induction Period (Maximum Increase) for the Question: "Do You Like the Drug?"
Description: as for outcome 10
Time Frame: End of Induction: 47.5 hours after first administration Peak Post Induction: Days 3-5
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sublingual Buprenorphine Soluble Film | Sublingual Buprenorphine/Naloxone Soluble Film
Number analyzed (Participants) | 18 | 16
units on a scale
  End of Induction | 14.9 (29.6) | 24.3 (37.0)
  Peak Post Induction | 61.7 (41.0) | 55.4 (35.8)
Statistical Analysis 1: Comparison: Sublingual Buprenorphine Soluble Film vs Sublingual Buprenorphine/Naloxone Soluble Film; Test type: Superiority or Other; p < 0.0001, Repeated measures model — The p-value was not adjusted for multiple comparisons; Group by time repeated measures model with a first-order autoregressive covariance structure

17. Secondary Outcome: Visual Analog Scale (VAS) Scores at End of Induction Period and the Post-induction Period (Maximum Increase) for the Question: "Does the Drug Make You Sick?"
Description: as for outcome 11
Time Frame: End of Induction: 47.5 hours after first administration Peak Post Induction: Days 3-5
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sublingual Buprenorphine Soluble Film | Sublingual Buprenorphine/Naloxone Soluble Film
Number analyzed (Participants) | 18 | 16
units on a scale
  End of Induction | 0 (0) | 0.3 (0.7)
  Peak Post Induction | 0 (0) | 0.7 (1.6)
Statistical Analysis 1: Comparison: Sublingual Buprenorphine Soluble Film vs Sublingual Buprenorphine/Naloxone Soluble Film; Test type: Superiority or Other; p = 0.238, Repeated measures model — The p-value was not adjusted for multiple comparisons; Group by time repeated measures model with a first-order autoregressive covariance structure

18. Secondary Outcome: Summary of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: Treatment-emergent AEs were defined as those starting on the day of the first treatment with buprenorphine soluble films or buprenorphine/ naloxone soluble films until residential research facility release, which typically happened on Day 6.
  Severity was graded by the investigator as mild (grade 1), moderate (grade 2) and severe (grade 3).
Time Frame: Day 1-6
Population: The randomized population included all subjects who were randomized to soluble films and received at least one dose of soluble films.
Measure: Number; unit: participants
Arm/Group | Sublingual Buprenorphine Soluble Film | Sublingual Buprenorphine/Naloxone Soluble Film
Number analyzed (Participants) | 20 | 18
participants
  With any TEAE | 20 | 18
  With grade 1 TEAE | 15 | 16
  With grade 2 TEAE | 19 | 16
  With grade 3 TEAE | 0 | 0

ADVERSE EVENTS:
Time Frame: Days 1-6. Treatment-emergent AEs were defined as those starting on the day of the first treatment with buprenorphine soluble films or buprenorphine/ naloxone soluble films until residential research facility release, which typically happened on Day 6.
Description: Adverse event data were collected by the investigator during daily subject interviews.
Arm/Group | Sublingual Buprenorphine Soluble Film | Sublingual Buprenorphine/Naloxone Soluble Film
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/18
Other Adverse Events (participants affected / at risk) | 20/20 | 18/18
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sublingual Buprenorphine Soluble Film (N=20) | Sublingual Buprenorphine/Naloxone Soluble Film (N=18)
Tachycardia (Cardiac disorders) | 6 | 3
Lacrimation increased (Ear and labyrinth disorders) | 4 | 5
Abdominal pain (Gastrointestinal disorders) | 1 | 3
Constipation (Gastrointestinal disorders) | 5 | 6
Dental caries (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 3 | 0
Dyspepsia (Gastrointestinal disorders) | 2 | 4
Nausea (Gastrointestinal disorders) | 6 | 5
Stomach discomfort (Gastrointestinal disorders) | 9 | 9
Toothache (Gastrointestinal disorders) | 2 | 1
Vomiting (Gastrointestinal disorders) | 2 | 3
Chills (General disorders) | 2 | 2
Cold sweat (General disorders) | 6 | 5
Hot flush (General disorders) | 0 | 2
Injection site erythema (General disorders) | 0 | 1 — Injection site AEs were due to morphine injections.
Injection site pruritus (General disorders) | 0 | 1 — Injection site AEs were due to morphine injections.
Irritability (General disorders) | 5 | 7
Fungal infection (Infections and infestations) | 0 | 1
Joint abscess (Infections and infestations) | 0 | 1
Liver function test abnormal (Investigations) | 0 | 1
Tuberculosis skin test positive (Investigations) | 3 | 1
Abscess limb (Musculoskeletal and connective tissue disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 | 1
Dizziness (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 11 | 10
Restlessness (Nervous system disorders) | 9 | 8
Tremor (Nervous system disorders) | 5 | 2
Anxiety (Psychiatric disorders) | 9 | 11
Drug withdrawal syndrome (Psychiatric disorders) | 14 | 13
Hyperventilation (Psychiatric disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 13 | 12
Dysuria (Renal and urinary disorders) | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 10 | 6
Yawning (Respiratory, thoracic and mediastinal disorders) | 4 | 4
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1
Piloerection (Skin and subcutaneous tissue disorders) | 2 | 7
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1
Tinea pedis (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 2 | 0
Hypertension (Vascular disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Proposed publications shall be submitted to Sponsor 30 days prior to submission for publication, and may be withheld for an additional period, up to 90 days, to allow Sponsor to file patent applications. If a multi-center publication isn't submitted for publication within 12 months of the conclusion of the Study at all sites, or is published in a shorter period, the results from the institution's site may be published individually.